CLINICAL TRIAL: NCT03773432
Title: Factors That Determine the Responses to Meal Ingestion: Meal Schedule and Gender Differences
Brief Title: Influence of Meal Schedule: Gender Differences
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PR(AG)338/2016G
Record Dates: First submitted 2018-12-05; First posted 2018-12-12 (Actual); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: Healthy
Keywords: meal ingestion; meal schedule; postprandial responses; hedonic sensations; homeostatic sensations

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Men (Other): In two separate days a probe meal (290 stewed beans, 35 g bread, 100 mL water; 549 Kcal) will be served at conventional and unconventional time.
  Interventions: Other: Probe meal
- Women (Other): In two separate days a probe meal (290 stewed beans, 35 g bread, 100 mL water; 549 Kcal) will be served at conventional and unconventional time.
  Interventions: Other: Probe meal

INTERVENTIONS:
Other: Probe meal — The probe meal will be administered either in the afternoon (conventional schedule) or in the morning (unconventional schedule).

SUMMARY:
Gender differences in the effect of meal schedule will be studied in a parallel design (10 women and 10 men). In two separate days a probe meal (290 stewed beans, 35 g bread, 100 mL water; 549 Kcal) will be administered in the afternoon, i.e. conventional schedule, and in the morning, i.e. unconventional schedule. The effect of meal schedule will be measured as the differences between the responses on both study days. Participants will be instructed to eat standard dinner the day before and to consume standard breakfast at home the day of the afternoon test. Studies will be conducted in a quiet, isolated room with participants siting on a chair. Perception will be measured at 5 min intervals 10 min before and 20 min after ingestion and at 10 min intervals up to 60 min after the probe meal.

ELIGIBILITY:
Inclusion Criteria:

* non-obese

Exclusion Criteria:

* history of gastrointestinal symptoms
* prior obesity
* use of medications
* history of anosmia and ageusia
* current dieting
* alcohol abuse
* psychological disorders
* eating disorders

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 20 (Actual)
Dates: Start 2018-08-13 (Actual); Primary Completion 2018-11-16 (Actual); Study Completion 2018-12-04 (Actual)

PRIMARY OUTCOMES:
Change in digestive well-being induced by meal schedule | 1 day
  Change in digestive well-being measured by a 10 cm scale graded from -5 (extremely unpleasant sensation) to +5 (extremely pleasant sensation) in response to afternoon and morning meals by repeated measures ANCOVA.

SECONDARY OUTCOMES:
Change in fullness sensation induced by meal schedule | 1 day
  Change in digestive well-being measured by a 10 cm scale graded from 0 (not at all) to 10 (very much) in response to afternoon and morning meals by repeated measures ANCOVA.
Change in mood induced by meal schedule | 1 day
  Change in mood measured by a 10 cm scale graded from -5 (negative) to +5 (positive) in response to afternoon and morning meals by repeated measures ANCOVA.
Change in hunger/satiety induced by meal schedule | 1 day
  Change in mood measured by a 10 cm scale graded from -5 (extremely hungry) to +5 (completely satiate) in response to afternoon and morning meals by repeated measures ANCOVA.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Vall d'Hebron, Barcelona, Spain

REFERENCES:
- [Background] Pribic T, Azpiroz F. Biogastronomy: Factors that determine the biological response to meal ingestion. Neurogastroenterol Motil. 2018 Jul;30(7):e13309. doi: 10.1111/nmo.13309. Epub 2018 Feb 2. PMID 29392797